CLINICAL TRIAL: NCT06943144
Title: Comparative Effects of Dual Task Training and Embodied Learning on Dual Task Performance in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/24/0735
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; Motor Coordination; Motor Skills; Psychomotor Performance; Cognitive Dysfunction
MeSH Terms: conditions — Down Syndrome; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be referred by Civil Hospital Sialkot and screened for eligibility. Guardians of eligible participants will provide informed consent prior to enrollment. A total of 22 participants will be randomly assigned via computer-generated randomization into two groups: Group A (Dual Task Learning) and Group B (Embodied Learning), with 11 participants in each. This single-blinded study will ensure the outcome assessor remains unaware of group assignments. Group A will engage in dual-task training-such as walking while solving math problems or identifying objects-twice a week for 30 minutes to improve cognitive-motor coordination. Group B will participate in embodied learning activities-such as yoga, gesture-based learning, storytelling, art, and sensory play-twice a week for 45-60 minutes to promote cognitive development through full-body engagement.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual task Training (Active Comparator): dual-task training, participants walk while doing cognitive tasks like counting or object identification to improve coordination and focus. Sessions are 30 minutes, twice weekly, with varying task difficulty and breaks for rest.
  Interventions: Other: Dual task Training
- Embodied Learning (Active Comparator): Participants attend twice-weekly 45-60 minute sessions using movement-based activities like yoga, art, and storytelling to enhance learning. Activities are tailored to individual needs.
  Interventions: Other: Embodied Learning

INTERVENTIONS:
Other: Dual task Training — In dual-task training, participants walk while performing cognitive tasks such as object identification, counting backward, or solving math problems. These exercises aim to improve coordination, attentional control, and dual-task performance by simultaneously engaging cognitive and motor functions. Training sessions are held twice a week, each lasting 30 minutes with breaks for rest and reflection. Tasks vary in complexity to progressively challenge participants and enhance both cognitive processing and gait stability.
  Arms: Dual task Training
Other: Embodied Learning — Participants in the embodied learning group engage in activities such as yoga, painting, sensory play, physical storytelling, gesture-based learning, and creative storytelling. These exercises use full-body movement to support learning and cognitive development. Examples include using gestures to reinforce concepts, acting out stories to blend movement with narrative, and engaging in yoga for focus and calmness. Art and sensory activities further promote creativity and tactile exploration. Sessions are held twice a week, lasting 45 to 60 minutes, and are tailored to individual needs and progress.
  Arms: Embodied Learning

SUMMARY:
This study aims to compare the effectiveness of embodied learning and dual-task training in improving coordination and cognitive function in children with Down syndrome. It involves 22 participants aged 7-12, excluding those with other neurological or orthopedic conditions. Participants will be referred from civil hospital Sialkot. Assessments include the Pediatric Balance Scale, Timed Up and Go Test, and other balance measures. Interventions include embodied learning (e.g., yoga, storytelling, sensory play) and dual-task activities (e.g., walking while solving puzzles). The goal is to enhance daily functioning and quality of life.

DETAILED DESCRIPTION:
Down Syndrome is Caused by an extra copy of chromosome 21, characterized by impaired motor skills, especially difficulties with coordination, and cognitive impairment. Improving these abilities is essential to raising the affected children's quality of life and everyday functioning. Dual task learning and embodied learning stand out among other interventions as effective strategies. While embodied learning uses physical motions to support cognitive growth, dual task learning mixes motor and cognitive tasks concurrently, testing the brain's capacity for multitasking. The purpose of this study is to compare how well embodied learning and dual task training work to improve dual task performance in kids with Down syndrome.

This study contains 22 participants age 7 to12 years and excludes participants with other neurological or orthopedic disorders, is focused on individuals who match the inclusion criteria Children that are being able to follow instructions. The Participants will be Referred by Civil hospital Sialkot. To test changes in motor coordination and balance, assessment tools such as the Pediatric Balance Scale (PBS), timed Up and Go Test, Single Leg Stance Test, Four Stage Balance Test, and 30-second Sit to Stand Test will be used. In order to evaluate cognitive engagement and the development of motor skills, dual task training setups (such as walking while labelling objects or balancing while solving puzzles) as well as embodied learning activities (such as Gesture-Based Learning, Physical Storytelling, Yoga, and Sensory Play Art) will be used. The purpose of this research is to offer useful knowledge about the effectiveness and practicality of various interventions in improving the everyday functioning and quality of life of children with Down syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with Down Syndrome
* Age 7 to 12 years
* Ability to follow instructions effectively

Exclusion Criteria:

* Neurological conditions (cerebral palsy or epilepsy)
* Orthopedic conditions (Foot Abnormalities,s Hip Dysplasia)
* Significant sensory impairments (e.g., severe hearing or vision impairments.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale(PBS) | 8 weeks
  The Pediatric Balance Scale (PBS) is a reliable and valid tool used to assess functional balance in school-aged children with mild to moderate motor impairments. It includes 14 items scored from 0 to 4, with a maximum score of 56. The PBS has shown excellent test-retest and interrater reliability and demonstrates strong correlations with functional outcomes such as self-care and mobility. It is also supported by its alignment with other motor assessments, making it an effective measure for evaluating and tracking balance skills in children with motor challenges.
Timed Up and Go (TUG) | 8 weeks
  The Timed Up and Go (TUG) test is a reliable and widely used tool for assessing mobility and fall risk across various populations. It demonstrates strong inter-rater and test-retest reliability, particularly in individuals with joint conditions. The test correlates well with key functional measures such as gait speed, postural control, and step length, and effectively predicts fall risk, making it a valuable tool for evaluating functional mobility.
Single Leg Stance (SLS) | 8 weeks
  The Single Leg Stance (SLS) Test evaluates static balance by measuring how long an individual can stand on one leg with eyes open and hands on hips. It is useful for detecting balance impairments, particularly in conditions like Total Knee Arthroplasty and Hip Osteoarthritis, and can indicate fall risk in older adults. The test demonstrates good reliability in these populations, though normative data remains limited.
30-Second Sit to Stand Test (30CST) | 8 weeks
  The 30-Second Sit to Stand Test (30CST) is a reliable and valid tool for assessing lower limb strength and endurance in diverse populations. It shows excellent test-retest, inter-rater, and intra-rater reliability, with strong correlations to other measures of lower extremity function, such as leg press performance. Widely used in clinical and research settings, the 30CST offers a consistent and objective measure of physical performance and functional capacity.
Four Stage Balance Test | 8 weeks
  The Four Stage Balance Test is reliable (interclass correlation = 0.66) over a 3-4-month interval with 187 subjects, indicating stable results. It demonstrates robust validity through strong correlations with established balance measures, making it an effective tool for identifying fall risk in older adults and guiding targeted interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Mahmood, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Izquierdo-Gomez R, Esteban-Cornejo I, Cabanas-Sanchez V, Marcos A, Gomez-Martinez S, Castro-Pinero J, Veiga OL; UP&DOWN Study Group. Are obesity and physical fitness associated with cardiovascular disease risk in adolescents with Down syndrome? The longitudinal UP&DOWN study. J Intellect Dev Disabil. 2023 Sep;48(3):247-259. doi: 10.3109/13668250.2023.2188876. Epub 2023 Mar 30. PMID 39815918